CLINICAL TRIAL: NCT07063810
Title: NEO-REEDUC - Mixed Reality for Motor Rehabilitation: a Prospective, Multicenter, Controlled, Randomized, Open Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Slb Pharma (Other)
Collaborators: Université de Caen Normandie (Other); NeoXpériences, Carpiquet, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEO-REEDUC
Record Dates: First submitted 2025-06-20; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Neurological Conditions; Brain Diseases; Cerebral Palsy; Parkinson Disease (PD); Multiple Sclerosis; Head Trauma; Ischemic Stroke; Cerebral Anoxia
Keywords: Mixed Reality; Neurological Conditions; Motor Rehabilitation; Postural Stability; Upper Limb; Locomotion
MeSH Terms: conditions — Brain Diseases; Cerebral Palsy; Parkinson Disease; Multiple Sclerosis; Craniocerebral Trauma; Ischemic Stroke; Hypoxia, Brain

STUDY DESIGN:
Intervention Model Description: A multicenter randomized controlled trial will be implemented across five different locations. One hundred and twenty patients will be randomly divided into an experimental group that will follow a mixed reality rehabilitation protocol with a pre-test and two post-test phases, with three weekly sessions for four weeks. A control group will only carry out the pre- and post-tests, and will perform their usual motor rehabilitation program.
Who Masked: Outcomes Assessor
Masking Description: The care providers will perform the 4-week rehabilitation program for the experimental group. The outcome assessors will only be in charge of the pre and post-test phases, and will not be informed on which group each participant was assigned to. All participants will receive a pseudonym which provides no information on their respective group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed Reality Group (Experimental): Patients will receive a mixed reality rehabilitation protocol for 4 weeks, on the basis of 3 sessions per week. These sessions will replace up to 3 usual motor rehabilitation sessions in order to limit any major increase in motor solicitations during this period.
  Interventions: Device: Mixed Reality Rehabilitation
- Control Group (No Intervention): Patients who will be assigned to the control group will follow their usual care for 4 weeks (usual motor activity, including rehabilitation and sports or physical activities). The rehabilitation protocol will be proposed after the second post-test phase.

INTERVENTIONS:
Device: Mixed Reality Rehabilitation — The mixed reality protocol will be based on 5 perceptual-motor activities (i.e., games specifically developed for the purposes of this study). The activities consist in walking to collect objects, avoid obstacles, or move the upper limbs to catch virtual balls or fit in narrow shapes.
  Three games will be performed per session, for a duration of 15 minutes each over 1h sessions with rest times.
  The level of the activities will be adapted to the performance of the participants during the course of the protocol, by manipulating game settings: necessary speed, accuracy and movement frequency.
  Arms: Mixed Reality Group

SUMMARY:
This study aims to assess the effectiveness of a motor rehabilitation protocol that includes mixed reality activities, compared to conventional rehabilitation, on postural stability in children and adult patients with neurological impairments.

DETAILED DESCRIPTION:
Conventional motor rehabilitation techniques applied to postural stability, locomotion or the upper limbs suffer from certain limitations. Studies in this field have highlighted the length and repetitiveness of these programs, which can lead to patient fatigue and pain. Combined with the lack of recreation and ecology in conventional therapies, which are often decontextualized and highly simplified, all these factors contribute to the lack of transposition of the improvements obtained into daily life activities (DLAs).

For several years now, the use of virtual reality (VR) and mixed reality (MR) have emerged as one of the most interesting solutions for overcoming these limitations. These technologies enable patients to take part in rehabilitation protocols under more controlled, progressive and attractive conditions, encouraging better patient adherence. These aspects guarantee effective rehabilitation and generalization of benefits to DLAs. In addition, they involve visuomotor coordination (skills involving the coordination of movements of different body segments with visual information previously perceived during execution), which is a cognitive ability widely transposable to DLAs.

Although some previous studies have investigated the effects of VR for motor rehabilitation, this technology also presents practical limitations related to the discomfort induced by the head-mounted displays (cybersickness, and physical discomforts caused by the weight of the display). Moreover, the use of VR tends to isolate the patient from their environment and therefore limits interaction with practitioners. Nevertheless, findings have shown the benefits of a VR protocol applied to motor rehabilitation in children and teenagers with cerebral palsy. The accuracy precision and fluidity of upper limb movements was improved, and the adherence to the protocol was strong.

In the line of these findings, the present protocol has several objectives: (1) to use MR, which seems to offer more possibilities while avoiding the disadvantages associated with VR, (2) to extend the applications of the proposed virtual rehabilitation tasks to other major motor functions - postural stability and locomotion as additional targets - and (3) to deploy these new rehabilitation methods to other patients likely to benefit from them (i.e. those with a functional disorder of neurological origin affecting their motor skills).

This study will include 120 patients with motor deficiencies of neurological origin, who will be randomly divided into two groups: one group receiving three weekly mixed reality rehabilitation sessions for four weeks, and a control group only following its usual care in the same period. Participants will be randomly matched for pathology, postural stability scores, age and sex. The effectiveness of the rehabilitation protocol will be evaluated through several clinical indicators of postural stability, locomotion and limb mobility as well as psychometrical measurements of fatigue, pain, motivation and quality of life.

ELIGIBILITY:
Inclusion Criteria:

- Adult patient (18 years old or older) with motor disorders related to a deficit in postural stability (mini-BESTest ≤ 25) which may be associated with a deficit in the use of upper limbs and locomotion, consecutive to : 1) either acquired neurological impairments (ischemic or hemorrhagic stroke in sub-acute or chronic phase, head trauma, benign tumor operated on with complete removal, cerebral anoxia) , or 2) a neurodegenerative affection (Parkinson's disease, Multiple Sclerosis).

OR

* Child or teenager patient (6 to 17 years old) with motor disorders related to a deficit in postural stability (mini-BESTest ≤ 25) which may be associated with a deficit in the use of upper limbs and locomotion, consecutive to 1) either spastic, dyskinetic or ataxic cerebral palsy, or 2) a similar impairment without diagnosis or of another etiology.
* Patient able to walk with or without technical aids and to perform voluntary upper limb movements.
* Patient able to understand and follow instructions or adapted communication.
* Patient having given written informed consent concerning his/her participation in the protocol OR (for children) whose parents have given their written informed consent.
* Patient covered by social security.

Exclusion Criteria:

* Patient with a severe intellectual disability.
* Patient with a severe attention deficit disorder.
* Patient whose epilepsy is not stable.
* Patient with pain preventing participation in the intended tasks of the protocol.
* Patient with an illness, medical condition or treatment incompatible with participation in the protocol.
* Patient with multiple sclerosis with relapse less than 3 months old.
* Simultaneous participation in other interventional research (1) that may exclude participation in the present study or (2) for which the exclusion period has not ended and whose nature may possibly impact the results of the present research.

In addition, the vulnerable persons mentioned in Articles L. 1121-5, L.1121-6 and L.1121-8 of the French Public Health Code are excluded from the study:

* Pregnant, nursing or parturient women.
* Persons deprived of their liberty by judicial or administrative decision, hospitalized without consent or admitted to a health or social institution for purposes other than research.
* Adults under legal protection or unable to express their consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in postural stability measured by the Mini-BesTest (or Kids Mini-BesTest) for children. | Pre-test (week 1), post-test (week 6) and 2-month follow-up (week 14).
  The test measures 5 aspects of postural stability in static and dynamic configurations over 14 items. Scores range from 0 to 28. A higher score indicates an overall better postural stability.

SECONDARY OUTCOMES:
Change in postural stability measured by the Functional Reach Test. | Pre-test (week 1), post-test (week 6) and 2-month follow-up (week 14).
  The test measures the maximum amplitude of a forward-reach movement before losing balance (in cm). A higher score means better performance .
Change in locomotor ability measured by the 6-minute walk test (6MWT) and the 10-meter walk test (10MWT). | Pre-test (week 1), post-test (week 6) and 2-month follow-up (week 14).
  The 6MWT measures the distance covered during a 6-minute period at a normal speed (in meters). The 10MWT measures the time (in seconds) taken to walk 10 meters at a fast speed.
Change in limb mobility measured by goniometry and a specific task implemented in the Mixed reality system. | Pre-test (week 1), post-test (week 6) and 2-month follow-up (week 14).
  Goniometry measures will be performed in an active rather than passive mode, in a standing position. The amplitude (in °deg) between a neutral position and the maximum movement will be measured on both shoulders, elbows, hips, knees and ankles when possible. The amplitude between a neutral station.
  The Mixed reality limb mobility task consists of 4 movements for each upper limb, and 3 movements for each lower limb, covering all dimensions. Joint amplitudes in °deg and percentage of maximum amplitude will be measured. Stride lengths front, back and sideways will also be computed during this task for each leg.
Change in quality of life measured by the MHAVIE questionnaire (measure of life habits). | Pre-test (week 1), post-test (week 6) and 2-month follow-up (week 14).
  The MHAVIE is a standard quality of life questionnaire validated in French-speaking populations. Participants (with or without help) indicate whether they are able to perform specific actions and if so, if they need technical or human help, as well as their level of satisfaction regarding their ability In the context of this study, 5 dimensions will be considered : locomotion, physical condition and psychological well-being, home, interpersonal relationships and leisure (total : 44 items maximum).
Change in pain, fatigue and motivation during the rehabilitation | Once at the beginning of the rehabilitation period (week 2) and once at the end of each week until the end of this period (weeks 2 to 5).
  Pain will be measured using the faces pain scale -revised, which is an illustrated 10-point scale.
  Fatigue will be measured by a 10-point Likert scale. Motivation will be measured using the Intrinsic motivation inventory. 12 questions will be asked, which patients will answer by rating on scales ranging from 1 to 7.
Change in cinematic parameters of upper limb movements and locomotion during the virtual activities (experimental group only). | For each trial of every virtual activity during the rehabilitation phase (weeks 2 to 5).
  Cinematic parameters of movements will be computed thanks to body tracking data recorded by the mixed reality device.Movement speed of the limbs and center of mass, as well as joint amplitudes during each trial of the virtual activities will be measured. The mixed reality activities can be performed in levels ranging from 1 to 10.
Progression in difficulty levels of the virtual activities (experimental group only). | For each trial of every virtual activity during the rehabilitation phase (weeks 2 to 5).
  The mixed reality activities can be performed in levels ranging from 1 to 10.
User experience measures as perceived by the care providers involved in the mixed reality rehabilitation protocol, using the AttrakDiff, UEQ and meCUE questionnaires. | At one point during the rehabilitation phase (during week 4 or 5).
  The AttrakDiff is a 28-item questionnaire. The care providers will rate the mixed reality system on 7-point scales delimited by pairs of opposite words. Measured dimensions are related to the pragmatic and hedonic quality of the system.
  the UEQ follows the same structure as the AttrakDiff and contains 26 items. The measured dimensions are attractiveness, perspicuity, efficiency, dependability, stimulation and novelty.
  The meCUE is a 30-item questionnaire (in its French version) questioning the several dimensions regarding the perception of the system, the positive and negative emotions during its use, and its consequences for future use intentions. Each item (except 1) is a 7-point Likert scale. The last item is a general appreciation of the system, on a 11-point scale ranging from -5 to +5.

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Continuing care and rehabilitation center (SSR) Les Monts d'Aunay, Aunay-sur-Odon, Normandy
  - Institute of Motor Education (IEM) François Xavier Falala, Hérouville-Saint-Clair, Normandy
  - Physical Medicine and Rehabilitation Center (CMPR) for Children and Adolescents La Clairière, Hérouville-Saint-Clair, Normandy
  - Physical Medicine and Rehabilitation Institute (IMPR) du bois de Lébisey, Hérouville-Saint-Clair, Normandy
  - La Musse Hospital, Saint-Sébastien-de-Morsent, Normandy

IPD SHARING:
Plan to Share IPD: No